CLINICAL TRIAL: NCT00857649
Title: A Randomised, Double-Blind, Parallel-Group Study Examining the Efficacy and Safety of Memantine in Patients With Moderate to Severe Dementia of the Alzheimer's Type
Brief Title: Efficacy and Safety of Memantine in Moderate to Severe Alzheimer's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10158
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Results first posted 2012-01-09 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-11

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Memantine (Experimental)
  Interventions: Drug: Memantine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine — 20 mg Oral Tablets Once Daily
  Other Names: Ebixa®
  Arms: Memantine
Drug: Placebo — Oral Tablets Once Daily
  Arms: Placebo

SUMMARY:
The primary objective of this study is to examine the efficacy of memantine on cognition and behavioural symptoms in outpatients with moderate to severe dementia of the Alzheimer's type.

DETAILED DESCRIPTION:
Memantine is a moderate affinity, uncompetitive N-methyl-D-aspartate (NMDA) receptor antagonist. Pre-clinical studies have demonstrated that memantine can decrease the neuronal toxicity associated with excessive glutamate release and calcium overload in neurons. Results from clinical trials in patients with moderate to severe Alzheimer's Disease (AD) have demonstrated memantine's efficacy and safety by showing positive treatment effects on cognitive, global and functional decline.

This 24-week randomised, double-blind, placebo-controlled, multicentre study examines the effect of memantine 20 mg, administered once daily, on cognitive and behavioural symptoms in outpatients diagnosed with moderate to severe AD and significant psychopathology.

ELIGIBILITY:
Inclusion Criteria:

Outpatients who:

* had a primary diagnosis of probable Alzheimer's Disease (AD) according to National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINDS-ADRDA) criteria, and with Diagnostic and Statistical Manual of Mental Disorders, 4th edition, text revised (DSM IV TR) criteria for dementia of the Alzheimer's type
* had moderate to severe dementia, defined as a Mini Mental State Examination (MMSE) total score >=5 and <=15 at screening. Before substantial protocol amendment SA04 (dated 7 October 2004) was implemented, the MMSE total score range at screening was >=8 and <=18. Substantial protocol amendment SA07 (dated 4 September 2009) allowed patients who had previously had an MMSE score of 16 or 17 to be re-screened >6 months after their initial screening and, if there was documented evidence of cognitive decline, to be enrolled in the study
* had a Neuropsychiatric Inventory (NPI) total score >=13 and an NPI agitation/aggression subitem score >=1 at screening and baseline
* did not have vascular dementia or a modified Hachinski Ischaemia Scale score >4 at screening

Exclusion Criteria:

* Evidence of clinically significant active disease, evidence of other neurological disorders, and previous treatment with memantine

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2003-12; Primary Completion 2010-04 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (23):
- Canada (23):
  - CA019, Edmonton, Alberta
  - CA033, Kelowna, British Columbia
  - CA034, Winnipeg, Manitoba
  - CA022, Saint John, New Brunswick
  - CA046, Kentville, Nova Scotia
  - CA045, Pictou, Nova Scotia
  - CA032, Burlington, Ontario
  - CA029, Orangeville, Ontario
  - CA004, Ottawa, Ontario
  - CA038, Peterborough, Ontario
  - CA009, Toronto, Ontario
  - CA037, Windsor, Ontario
  - CA005, Beauport, Quebec
  - CA023, Greenfield Park, Quebec
  - CA013, Montreal, Quebec
  - CA031, Sherbrooke, Quebec
  - CA012, Sherbrooke, Quebec
  - CA030, Vanier, Quebec
  - CA017, Verdun, Quebec
  - CA015, Regina, Saskatchewan
  - CA040, Saskatoon, Saskatchewan
  - CA043, Kelowna
  - CA042, Penticton

REFERENCES:
- [Result] Herrmann N, Gauthier S, Boneva N, Lemming OM; 10158 Investigators. A randomized, double-blind, placebo-controlled trial of memantine in a behaviorally enriched sample of patients with moderate-to-severe Alzheimer's disease. Int Psychogeriatr. 2013 Jun;25(6):919-27. doi: 10.1017/S1041610213000239. Epub 2013 Mar 8. PMID 23472619

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients were recruited from the investigators' outpatient clinics.
Pre-assignment Details: At the Baseline Visit, the patients were randomised (1:1) to 24 weeks of treatment with placebo or memantine. Patients randomised to memantine were up-titrated in weekly increments of 5 mg over a 4-week dose-escalation period. The target dose of 20 mg/day was administered at the start of the fourth week and maintained for the rest of the study.
Period: Overall Study
Arm/Group | Memantine | Placebo
Started | 182 | 187
Completed | 151 | 155
Not Completed | 31 | 32
Not completed — Adverse Event | 15 | 10
Not completed — Non-compliance | 1 | 1
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal of Consent | 10 | 7
Not completed — Nursing Home Placement | 2 | 9
Not completed — Other Reasons | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Memantine | Placebo | Total
Number analyzed (Participants) | 182 | 187 | 369
Age Continuous [Mean (Standard Deviation); unit: years] | 74.7 (7.9) | 75.1 (6.9) | 74.9 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 110 | 215
  Male | 77 | 77 | 154
NPI: Baseline Total Score [Mean (Standard Deviation); unit: Scores on a scale] — The Neuropsychiatric Inventory (NPI) is a validated scale that assesses behavioural disturbances in patients with dementia. The 12 item version consists of 10 behavioural and 2 neurovegetative areas. It provides both a total score as well as scores for a number of sub-scales. The frequency, severity and caregiver distress for each domain are measured. The NPI is based upon responses obtained from the caregiver. The total score is from 0 to 144. A higher score reflects more frequency and severity of the disturbances.
  Scores on a scale | 30.9 (14.8) | 29.2 (13.3) | 30.1 (14.0)
SIB: Baseline Total Score [Mean (Standard Deviation); unit: Scores on a scale] — The Severe Impairment Battery (SIB) is a validated scale used to assess cognitive function in patients with moderate to severe dementia. Items are single words or one-step commands combined with gestures. Nine domains are assessed, and the total score is between 0 and 100. A lower total score reflects the loss of cognitive function.
  Scores on a scale | 82.3 (14.6) | 82.0 (12.9) | 82.1 (13.7)
CIBIC-plus: Baseline Severity Score [Mean (Standard Deviation); unit: Scores on a scale] — The Clinician's Interview-Based Impression of Change-Plus Version (CIBIC-plus) is a global rating that is derived through an independent, comprehensive interview with the patient and caregiver by a rater who is barred from knowledge of all other psychometric test scores conducted as part of this protocol as well as from reported safety data. The rating is made on a 7-point scale ranging from "1 = marked improvement" to "7 = marked worsening". A score of "4" indicates no change.
  Scores on a scale | 4.4 (0.9) | 4.4 (0.9) | 4.4 (0.9)
ADCS-ADL - 19 items: Baseline Total Score [Mean (Standard Deviation); unit: Scores on a scale] — Alzheimer's Disease Cooperative Study - Activities of Daily Living Inventory (ADCS-ADL) - 19 items total score version for moderate to severe AD will measure patient's functioning. This battery of ADL questions is used here to measure the functional capabilities of patients with dementia. The inventory is done by interviewing a person in close contact with the patient and covers the most usual and consistent performance of the patient over the preceding 4 weeks. Total score is from 0 to 54. The higher score, the lower impairment.
  Scores on a scale | 35.3 (9.9) | 36.4 (8.6) | 35.8 (9.3)
CMAI - Long Form: Baseline Total Score [Mean (Standard Deviation); unit: Scores on a scale] — The Cohen-Mansfield Agitation Inventory (CMAI) - Long Form looks specifically at agitated behaviour in patients with cognitive impairment. It is a seven-point rating scale assessing the frequency of up to 29 agitated behaviours, ranging from "1 = Never" to "7 = Several times an hour". Rating is based on responses obtained from interviews with the caregiver. The total score ranges from 29 to 203, with a higher score reflecting more frequent behavioural disturbances.
  Scores on a scale | 46.8 (10.9) | 47.0 (10.9) | 46.9 (10.9)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Memantine on Behavioural Symptoms in Outpatients With Moderate to Severe Dementia of the Alzheimer's Type Using the NPI - 12 Items Version Total Score.
Description: Change from Baseline in Neuropsychiatric Inventory (NPI) total score.
  NPI is a validated scale that assesses behavioural disturbances in patients with dementia. The 12 item version consists of 10 behavioural and 2 neurovegetative areas. It provides both a total score as well as scores for a number of sub-scales. The frequency, severity and caregiver distress for each domain are measured. The NPI is based upon responses obtained from the caregiver. The total score is from 0 to 144. A higher score reflects more frequency and severity of the disturbances.
Time Frame: Baseline to Week 24
Population: Full-analysis Set (FAS) - all randomised patients on current treatment with an acetylcholinesterase inhibitor (AChEI) who took at least one dose of investigational medicinal product (IMP) and had at least one post-baseline assessment on both co-primary efficacy variables.
  Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 159 | 165
Scores on a scale | -3.90 (1.24) | -5.13 (1.23)
Statistical Analysis 1: Comparison: Memantine vs Placebo; Test type: Superiority or Other; p = 0.418, ANCOVA; Centre and treatment as factors and baseline score as covariate. Estimate based on Least Squares; Mean Difference (Final Values) = 1.23, 95% CI 2-sided [-1.75 to 4.21], Standard Error of Mean 1.52

2. Primary Outcome: Efficacy of Memantine on Cognition in Outpatients With Moderate to Severe Dementia of the Alzheimer's Type Using the SIB Total Score.
Description: Change from Baseline in Severe Impairment Battery (SIB) total score.
  SIB is a validated scale used to assess cognitive function in patients with moderate to severe dementia. Items are single words or one-step commands combined with gestures. Nine domains are assessed, and the total score is between 0 and 100. A lower total score reflects the loss of cognitive function.
Time Frame: Baseline to Week 24
Population: FAS; LOCF
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 159 | 165
Scores on a scale | -2.34 (0.76) | -1.86 (0.75)
Statistical Analysis 1: Comparison: Memantine vs Placebo; Test type: Superiority or Other; p = 0.603, ANCOVA; Centre and treatment as factors and baseline score as covariate. Estimate based on Least Squares; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-2.30 to 1.34], Standard Error of Mean 0.92

3. Secondary Outcome: Efficacy of Memantine on Global Condition Using CIBIC-plus.
Description: Clinician's Interview-Based Impression of Change-Plus Version (CIBIC-plus). Improvement evaluated with reference to Baseline.
  CIBIC-plus is a global rating that is derived through an independent, comprehensive interview with the patient and caregiver by a rater who is barred from knowledge of all other psychometric test scores conducted as part of this protocol as well as from reported safety data. The rating is made on a 7-point scale ranging from "1 = marked improvement" to "7 = marked worsening". A score of "4" indicates no change.
Time Frame: Baseline to Week 24
Population: FAS; Observed Cases (OC).
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 135 | 140
Scores on a scale | 4.68 (0.11) | 4.63 (0.11)
Statistical Analysis 1: Comparison: Memantine vs Placebo; Test type: Superiority or Other; p = 0.734, ANCOVA; Centre and treatment as factors and baseline score as covariate. Estimate based on Least Squares; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.22 to 0.31], Standard Error of Mean 0.13

4. Secondary Outcome: Efficacy of Memantine on Functioning Using ADCS-ADL - 19 Items Total Score.
Description: Change from Baseline on the Alzheimer's Disease Cooperative Study - Activities of Daily Living Inventory (ADCS-ADL) 19-item version total score.
  ADCS-ADL- 19 items version for moderate to severe AD will measure patient's functioning. This battery of ADL questions is used here to measure the functional capabilities of patients with dementia. The inventory is done by interviewing a person in close contact with the patient and covers the most usual and consistent performance of the patient over the preceding 4 weeks. Total score is from 0 to 54. The higher score, the lower impairment.
Time Frame: Baseline to Week 24
Population: FAS; OC
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 136 | 140
Scores on a scale | -4.36 (0.67) | -2.56 (0.65)
Statistical Analysis 1: Comparison: Memantine vs Placebo; Test type: Superiority or Other; p = 0.017, ANCOVA; Centre and treatment as factors and baseline score as covariate. Estimate based on Least Squares; Mean Difference (Final Values) = -1.80, 95% CI 2-sided [-3.29 to -0.32], Standard Error of Mean 0.75

5. Secondary Outcome: Efficacy of Memantine on Functioning Using CMAI - Long Form Total Score.
Description: Change from Baseline on the Cohen-Mansfield Agitation Inventory (CMAI) - Long Form total score.
  CMAI - Long Form looks specifically at agitated behaviour in patients with cognitive impairment. It is a seven-point rating scale assessing the frequency of up to 29 agitated behaviours, ranging from "1 = Never" to "7 = Several times an hour". Rating is based on responses obtained from interviews with the caregiver. The total score ranges from 29 to 203, with a higher score reflecting more frequent behavioural disturbances.
Time Frame: Baseline to Week 24
Population: FAS; OC
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 134 | 139
Scores on a scale | -0.26 (0.79) | -1.16 (0.79)
Statistical Analysis 1: Comparison: Memantine vs Placebo; Test type: Superiority or Other; p = 0.360, ANCOVA; Centre and treatment as factors and baseline score as covariate. Estimate based on Least Squares; Mean Difference (Final Values) = 0.90, 95% CI 2-sided [-1.03 to 2.83], Standard Error of Mean 0.98

ADVERSE EVENTS:
Time Frame: Up to 28 weeks
Arm/Group | Memantine | Placebo
Serious Adverse Events (participants affected / at risk) | 18/182 | 11/187
Other Adverse Events (participants affected / at risk) | 51/182 | 35/187
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Memantine (N=182) | Placebo (N=187)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Local swelling (General disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Acute sinusitis (Infections and infestations) | 1 | 0
Bronchitis viral (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 2 | 0
Viral infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Convulsion (Nervous system disorders) | 0 | 1
Dementia alzheimer's type (Nervous system disorders) | 0 | 1
Aggression (Psychiatric disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Hallucination, auditory (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Personality disorder (Psychiatric disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Social stay hospitalisation (Social circumstances) | 1 | 1
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Memantine (N=182) | Placebo (N=187)
Nausea (Gastrointestinal disorders) | 4 | 11
Fall (Injury, poisoning and procedural complications) | 19 | 8
Weight decreased (Investigations) | 11 | 5
Somnolence (Nervous system disorders) | 10 | 5
Agitation (Psychiatric disorders) | 15 | 7

LIMITATIONS AND CAVEATS:
Long recruitment, premature termination, substantial protocol changes; baseline imbalances (concomitant medication and severity of agitation). Variability across sites in reported events frequency (50% of agitation reports from a single site)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and H. Lundbeck A/S. Manuscripts and abstracts must be sent to H. Lundbeck A/S at least one month prior to submission for publication or presentation.